CLINICAL TRIAL: NCT03088397
Title: Effectiveness of a Patient Decision Aid in Immediate Postpartum Contraceptive Counseling
Acronym: POCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Erika Levi, Co-Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-6978
Record Dates: First submitted 2016-09-07; First posted 2017-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient decision aid (Experimental): Group receives the patient decision aid, POCO (POstpartum Contraceptive Options), a grid with various contraceptive options across the columns and characteristics of each option in rows. Group receives Shared Decision Making counseling afterwards.
  Interventions: Behavioral: Patient Decision Aid; Behavioral: Shared- Decision Making Counseling
- Website information (Active Comparator): Group receives directions on how to get to bedsider.org information pages regarding contraceptive choices. Group receives Shared Decision Making counseling afterwards.
  Interventions: Behavioral: Website; Behavioral: Shared- Decision Making Counseling
- Standard of care (Active Comparator): Group receives standard brochure on contraception in their postpartum packet. Group receives Shared Decision Making counseling afterwards.
  Interventions: Behavioral: Shared- Decision Making Counseling

INTERVENTIONS:
Behavioral: Patient Decision Aid — One sheet of postpartum contraceptive information arranged in a grid.
  Arms: Patient decision aid
Behavioral: Website — Patient directed to website with information on various contraceptive methods.
  Arms: Website information
Behavioral: Shared- Decision Making Counseling — Counseling using principles of shared-decision making

SUMMARY:
Effective physician-patient communication in postpartum contraceptive counseling is essential for patients to meet their contraceptive needs and reduce the risk of rapid repeat pregnancies. This project will utilize a patient decision aid to facilitate shared decision making in the immediate postpartum setting, assess the effectiveness of such aid in "decision quality" and "decision-making process quality", and observe its effects on contraceptive choice mix at the time of discharge.

DETAILED DESCRIPTION:
More than 51% of pregnancies in the US are unintentional. Of the unintended pregnancies, 43% are attributable to incorrect or inconsistent use of contraceptive methods. Gaps in contraceptive use can arise from a misalignment of the patient's needs or preferences and her chosen method. This is particularly salient in the postpartum setting; nearly two-thirds of women in their first year of postpartum have unmet need for family planning, and adolescents in particular are at high risk for repeat pregnancies within a year.

Effective physician-patient communication in postpartum contraceptive counseling is essential for patients to meet their contraceptive needs. Previously, there has been an emphasis on "informed choice" model for counseling, in which the clinician's role is to provide information to the patient in order to facilitate her choice of a contraceptive method. The provider does not actively participate in the process of selecting the method, in the spirit of respecting patient autonomy. Dehlendorf et al. has shown that while women do value autonomy in making a decision about their contraceptive method, they prefer more provider involvement in the decision making process than the "informed choice" model allows. This has given room for a rise in interest in Shared Decision Making (SDM) model of counseling for contraceptive care. In the SDM model, the clinical plays a supportive role in patient decision making, by not only providing information but also guiding the patient through her deliberation. While the final decision is left in the hands of the patient, they are given support to identify their preferences and needs, and to align them with an option that best matches her preferences and needs.

Various decision making tools have been developed to facilitate SDM. One method is to display all available options in one axis, and frequently-asked questions regarding each option in the other axis. Patients are asked to select frequently-asked questions that address their concerns, thereby sorting through the most pertinent information regarding their options in one view. Research has shown that such patient decision aids (PtDA) help patients understand their options, feel more informed, participate in decision making, and have more accurate expectations of possible outcomes.

The goal of this project is to utilize a PtDA to facilitate SDM in the immediate postpartum setting, assess the effectiveness of such PtDA on decision quality and decision-making process quality (as defined and measured by previously validated survey tools), and to observe its effects on patients' contraceptive choice at the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English or Spanish speaking
* Delivered during current admission to hospital
* Postpartum day 1 or post-op day 1 or 2

Exclusion Criteria:

* Females less than 14 years of age
* Status post sterilization or hysterectomy
* Received an intrauterine device immediately after delivery (postplacental)
* Does not have a smartphone capable of browsing the internet

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Quality of decision making process | 6 months
  Preparation for Decision Making scale

SECONDARY OUTCOMES:
Choice in Contraceptive Method | 6 months
  Data will be collected regarding which method of contraception each participant chooses to use

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finer LB, Zolna MR. Shifts in intended and unintended pregnancies in the United States, 2001-2008. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S43-8. doi: 10.2105/AJPH.2013.301416. Epub 2013 Dec 19. PMID 24354819
- [Background] Frost JJ, Darroch JE, Remez L. Improving contraceptive use in the United States. Issues Brief (Alan Guttmacher Inst). 2008;(1):1-8. PMID 18561392
- [Background] Donnelly KZ, Foster TC, Thompson R. What matters most? The content and concordance of patients' and providers' information priorities for contraceptive decision making. Contraception. 2014 Sep;90(3):280-7. doi: 10.1016/j.contraception.2014.04.012. Epub 2014 Apr 30. PMID 24863169
- [Background] Dehlendorf C, Levy K, Kelley A, Grumbach K, Steinauer J. Women's preferences for contraceptive counseling and decision making. Contraception. 2013 Aug;88(2):250-6. doi: 10.1016/j.contraception.2012.10.012. Epub 2012 Nov 21. PMID 23177265
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Stacey D, Bennett CL, Barry MJ, Col NF, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Legare F, Thomson R. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD001431. doi: 10.1002/14651858.CD001431.pub3. PMID 21975733
- [Background] Lopez LM, Grey TW, Chen M, Hiller JE. Strategies for improving postpartum contraceptive use: evidence from non-randomized studies. Cochrane Database Syst Rev. 2014 Nov 27;2014(11):CD011298. doi: 10.1002/14651858.CD011298.pub2. PMID 25429714
- [Background] Sepucha KR, Borkhoff CM, Lally J, Levin CA, Matlock DD, Ng CJ, Ropka ME, Stacey D, Joseph-Williams N, Wills CE, Thomson R. Establishing the effectiveness of patient decision aids: key constructs and measurement instruments. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S12. doi: 10.1186/1472-6947-13-S2-S12. Epub 2013 Nov 29. PMID 24625035